CLINICAL TRIAL: NCT03978767
Title: Preeclampsia And Nonsteroidal Drugs for Analgesia (PANDA): a Randomized Non Inferiority Trial
Brief Title: Preeclampsia And Nonsteroidal Drugs for Analgesia: a Randomized Non Inferiority Trial
Acronym: PANDA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201901202
Record Dates: First submitted 2019-05-18; First posted 2019-06-07 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Preeclampsia Severe; Preeclampsia Postpartum
Keywords: NSAIDs; Ibuprofen
MeSH Terms: interventions — Ibuprofen; Ketorolac; Acetaminophen; Oxycodone

STUDY DESIGN:
Intervention Model Description: Randomized non-inferiority clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NSAID Analgesic bundle (Experimental): Ibuprofen 600mg PO q 6 hrs as needed for pain, Acetaminophen 1000mg q 8 hrs as needed for pain, and Oxycodone 5 to 10 mg q 4 hrs as needed for pain. In patients undergoing cesarean section, ketorolac 30mg IV q 6 hrs may be substituted as an IV alternative to ibuprofen for the first 24 hours after surgery
  Interventions: Drug: Ibuprofen 600 mg; Drug: Ketorolac; Drug: Acetaminophen; Drug: Oxycodone
- NSAID free analgesic bundle (Active Comparator): Acetaminophen 1000mg q 8 hrs as needed for pain, and Oxycodone 5 to 10 mg q 4 hrs as needed for pain.
  Interventions: Drug: Acetaminophen; Drug: Oxycodone

INTERVENTIONS:
Drug: Ibuprofen 600 mg — NSAID pain medication to be used in the experimental bundle for postpartum analgesia
  Arms: NSAID Analgesic bundle
Drug: Ketorolac — NSAID analgesic to be used in the experimental bundle for postpartum analgesia in patients who underwent cesarean section
  Arms: NSAID Analgesic bundle
Drug: Acetaminophen — Analgesic medication to be used in both treatment arms
Drug: Oxycodone — Analgesic medication to be used in both treatment arms

SUMMARY:
A randomized non-inferiority trial of women with preeclampsia with severe features to determine if the addition of nonsteroidal anti-inflammatory drugs is inferior or non-inferior to standard analgesic bundles in their impact on postpartum hypertension.

DETAILED DESCRIPTION:
Recently published clinical guidelines for the care of women with hypertensive disorders recommended that nonsteroidal anti-inflammatory drugs (NSAIDs) should be withheld from patients with hypertension that persists for more than one day postpartum (1). This recommendation is based in data from the general medicine literature, which suggests a role of NSAIDs in precipitating hypertension in non-pregnant adults (2,3). It may also draw from previously published case reports of post-partum hypertension that were thought to be NSAID induced (4). There has been a paucity of data from the obstetric literature to support or rebuff this recommendation. As the opioid crisis worsens in the United States, additional attention and resources have focused on limiting the use of narcotic medications. The effective employment of non-opioid analgesics has been shown to reduce narcotic use (5). Ibuprofen and other NSAIDs are the most effective and most commonly prescribed analgesics for postpartum pain, but clinicians now find themselves stuck between these recommendations and their efforts to limit unnecessary opioid prescriptions.

The investigators propose a randomized controlled non-inferiority trial of women with preeclampsia comparing a postpartum analgesic protocol that includes NSAIDs, to one that excludes them. The central hypothesis is that NSAID use does not worsen hypertensive diseases of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women at > 23 weeks gestational age undergoing vaginal or cesarean delivery at Barnes-Jewish Hospital with:
* An antepartum diagnosis of preeclampsia with severe features
* Pre-eclampsia with severe features will be defined as:
* Elevated blood pressure ≥ 160/110, or
* Pre-eclampsia in the setting of thrombocytopenia (platelet count < 100,000), or
* Impaired liver function (AST elevated to twice upper limit of normal), or
* Persistent epigastric pain, or
* Renal insufficiency (serum creatinine of 1.1 mg/dl or doubling of prior value), or
* Pulmonary edema, or
* New onset visual disturbance or headache unresponsive to therapy.

Exclusion Criteria:

* NSAID allergy
* Allergy to acetaminophen
* Antihypertensive use in this pregnancy prior to 20 weeks gestation
* Chronic kidney disease or Acute kidney injury with Creatine clearance less than 60 mL/min
* Inability to obtain consent
* Opioid abuse disorder
* Peptic ulcer disease.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
postpartum antihypertensive requirements | at the end of hospitalization, up to 7 days after randomization
  measurement of anti-hypertensive requirements at time of discharge

SECONDARY OUTCOMES:
Postpartum pain scores | From randomization to 6 weeks after randomization
  Evaluate the effect of NSAIDs on patient perception of pain
Postpartum opioid use | From randomization to 6 weeks after randomization
  Compare the opioid requirements in each arm
Mean arterial blood pressure | From randomization to 6 weeks after randomization
  Compare peak, average and median MAPs postpartum
End organ damage | during hospitalization, an average of 4 days
  Evaluate for evidence of renal, hepatic or neurological injury in the poatpartum period
Hospital readmission | From randomization to 6 weeks after randomization
  Evaluate the incidence of hospital readmission rate postpartum
Continued anti-hypertensive requirement | up to 6 weeks
  evaluate the need for antihypertensive medications at 6 weeks postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Background] Lo JO, Mission JF, Caughey AB. Hypertensive disease of pregnancy and maternal mortality. Curr Opin Obstet Gynecol. 2013 Apr;25(2):124-32. doi: 10.1097/GCO.0b013e32835e0ef5. PMID 23403779
- [Background] Sibai B, Dekker G, Kupferminc M. Pre-eclampsia. Lancet. 2005 Feb 26-Mar 4;365(9461):785-99. doi: 10.1016/S0140-6736(05)17987-2. PMID 15733721
- [Background] Mogos MF, Salemi JL, Spooner KK, McFarlin BL, Salihu HH. Hypertensive disorders of pregnancy and postpartum readmission in the United States: national surveillance of the revolving door. J Hypertens. 2018 Mar;36(3):608-618. doi: 10.1097/HJH.0000000000001594. PMID 29045342
- [Background] Viteri OA, England JA, Alrais MA, Lash KA, Villegas MI, Ashimi Balogun OA, Chauhan SP, Sibai BM. Association of Nonsteroidal Antiinflammatory Drugs and Postpartum Hypertension in Women With Preeclampsia With Severe Features. Obstet Gynecol. 2017 Oct;130(4):830-835. doi: 10.1097/AOG.0000000000002247. PMID 28885417

DOCUMENTS (3):
  • Study Protocol (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT03978767/Prot_001.pdf
  • Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT03978767/SAP_000.pdf
  • Informed Consent Form (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT03978767/ICF_002.pdf